CLINICAL TRIAL: NCT06000215
Title: Credibility of Ultrasound Detection of Female Genital Prolapse Mesh
Acronym: KIDS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Edward Morcos, MD, PhD. Senior Consultant., Karolinska Institutet
Other Study IDs: Dnr: 2018/1523-31
Record Dates: First submitted 2023-02-16; First posted 2023-08-21 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Uphold™ Lite Vaginal mesh - Boston Scientific (Anterior): Patients previousely received the Uphold™ Lite for the surgical management of apical and/or anterior vaginal mesh prolapse.
  Interventions: Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners are blinded to each other and to the previous prolapse surgery.; Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners is now being informed of the previous prolapse surgery.
- Pinnacle posterior Vaginal mesh - Boston Scientific: Patients previousely received the Pinnacle posterior Vaginal mesh for the surgical management of posterior and/or apical vaginal mesh prolapse.
  Interventions: Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners are blinded to each other and to the previous prolapse surgery.; Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners is now being informed of the previous prolapse surgery.
- Artisyn® Y-Shaped Mesh (Robotic-assisted Sacral colpopexy): Patients previousely received the Artisyn® Y-Shaped Mesh via robotic-assisted approach Patients previousely received th Artisyn® Y-Shaped Mesh via robotic-assisted approach for the surgical management of apical prolapse..
  Interventions: Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners are blinded to each other and to the previous prolapse surgery.; Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners is now being informed of the previous prolapse surgery.
- Native tissue repair: Patients previousely received native tissue repair for the surgical management of prolapse.
  Interventions: Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners are blinded to each other and to the previous prolapse surgery.; Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners is now being informed of the previous prolapse surgery.

INTERVENTIONS:
Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners are blinded to each other and to the previous prolapse surgery. — Each examiner to answer:
  1. Is there a mesh or not: Yes or No
  2. If Yes:
     * Which type of mesh? Uphold, Pinnacle Posterior or Artisyn® Y-Shaped Mesh
     * What is the length of the mesh in a single midsagittal view image
  3. Examination record time is to be registered.
  Other Names: Vaginal ultrasound examination, two different examiners. The examiners are blinded to each other and to the previous prolapse surgery
Diagnostic Test: Perineal/introital ultrasound examination, two different examiners. The examiners is now being informed of the previous prolapse surgery. — Each examiner to answer:
  1. Is there a mesh or not: Yes or No
  2. If Yes:
     * Which type of mesh? Uphold, Pinnacle Posterior or Artisyn® Y-Shaped Mesh
     * What is the length of the mesh in a single midsagittal view image
  3. Examination record time is to be registered.
  Other Names: Vaginal ultrasound examination, two different examiners. The examiners is now being informed of the previous prolapse surgery.

SUMMARY:
The aim of the study is to investigate the credibility of ultrasound in detection of synthetic polypropylene vaginal implants. In detail, the study investigates if the ultrasound examiner experience and the standard method of examination may affect the detection of synthetic polypropylene vaginal implants by ultrasound.

The primary hypothesis is if 90% of prolapse mesh could be detected by the ultrasound examiners who are blinded to the previous prolapse surgery, the ultrasound is credible for prolapse mesh detection.

The secondary hypothesis is if the ultrasound detection is not significantly different between the ultrasound examiners, the method of ultrasound examination is mandatory to acheive credible ultrasound detection of the prolapse mesh.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a common condition in post-delivery and post-reproductive aged women (1). The lifetime risk of undergoing a single operation for prolapse or incontinence by age 80 is 11% (2). POP is mainly classified into three compartments: anterior, middle (apical) or posterior (1). Apical defects include descensus uteri or vaginal vault prolapse after previous hysterectomy. Traditional Surgical repairs of POP using native connective tissues are commonly used but the risk for POP recurrence is high if apical prolapse is present (ca 60%) (1). Thus, the development of different mesh types using different approaches to support the vaginal apex (uterus or vaginal top) is highly growing. Surgery may be done by transvaginal mesh (TVM) or robotic-assisted sacroclpopexy (3). Increasing evidence show effectivity of both methods and improved HR-QoL after surgery (4, 5, 6, 7, 8, 9). However, PFD including urinary incontinence, urinary bladder emptying disorders and prolapse recurrence may be postoperative conditions (1, 2).

Growing needs worldwide is to improve diagnostic methods such as ultrasonography (US). This may improve the clinical knowledge to be further used for management of pelvic floor disorders (PFD). US is a cheap and safe method as compared to magnetic resonance (MR) or computed tomography (CT) (10). Thus, if using US to provide clinical examination instead of MR and CT the health care cost may be reduced. Indeed, US can provide imaging in some cross sections giving same imaging results of MR (10).

Some studies have been investigating the use of endo-vaginal, trans-perineal/introital and trans-labial US techniques in detection of implants with more focus on TVT-surgery (Tension-free vaginal tape) for urinary incontinence (UI) and to some extent detection of prolapse mesh (11). However, sensitivity of depiction has been reported to 92% at rest and 72% on physical examination when using endovaginal US examination (11). Also, the depiction is dependent on the US expertise since no standardization has been achieved. Furthermore, the presence of scar tissues following previous POP or UI surgery in the pelvic floor region has been described as an interrupting factor for prediction (10).

Thus, development of a standardized US prediction of implants in order to elucidate anatomical and functional information in the pelvic floor when POP mesh is implanted may be useful in management of PFD. It is to investigate the sensitivity and reproducibility of this US model of examination.

The purpose of the present study is to investigate the credibility of the US detection of prolapse mesh implants when a standardized method of US examination is performed.

Methodology of the present study Perineal/introital and vaginal ultrasound examination is done using a standard protocol by two different US examiners of four groups of patients previously received prolapse surgery. Each examiner is to be entered from the pre-examination room, do all requested examinations in one time, and leave from the examination room to be followed by the next examiner without meeting each other. Thus, the ultrasound examiners are to be blinded to each other and to the previous prolapse surgery. A controller is appointed to introduce each examiner from the pre-examination room, record the time of each examination and collect the results of examinations. The statistician is also to be blinded to the group of examination.

References

1. Barber MD, Maher C. Apical prolapse. Int Urogynecol J. 2013; 24(11):1815-33.
2. Olsen AL, Smith VJ, Bergstrom JO, Colling JC, Clark AL. Epidemiology of surgically managed pelvic organ prolapse and urinary incontinence. Obstet Gynecol. 1997 Apr;89(4):501-6.
3. Maher C, Feiner B, Baessler K, Schmid C. Surgical management of pelvic organ prolapse in women. Cochrane Database Syst Rev. 2013 Apr 30;(4):CD004014.
4. Oliver JL, Kim JH. Robotic Sacrocolpopexy-Is It the Treatment of Choice for Advanced Apical Pelvic Organ Prolapse? Curr Urol Rep. 2017 Sep;18(9):66-74.
5. Rahkola-Soisalo P, Mikkola TS, Altman D, Falconer C; for Nordic TVM Group. Pelvic Organ Prolapse Repair Using the Uphold Vaginal Support System: 5-Year Follow-up. Female Pelvic Med Reconstr Surg. 2017 Dec 11. Fortcoming 2018.
6. Gutman RE, Rardin CR, Sokol ER, Matthews C, Park AJ, Iglesia CB, st al. Vaginal and laparoscopic mesh hysteropexy for uterovaginal prolapse: a parallel cohort study. Am J Obstet Gynecol. 2017. Jan;216(1):38.e1-38.e11.
7. Lua LL, Vicente ED, Pathak P, Lybbert D, Dandolu V. Comparative analysis of overall cost and rate of healthcare utilization among apical prolapse procedures. Int Urogynecol J. 2017 Oct;28(10):1481-8.
8. Rahkola-Soisalo P, Altman D, Falconer C, Morcos E, Rudnicki M, Mikkola TS. Quality of life after Uphold™ Vaginal Support System surgery for apical pelvic organ prolapse-A prospective multicenter study. Eur J Obstet Gynecol Reprod Biol. 2017 Jan;208:86-90. doi: 10.1016/j.ejogrb.2016.11.011. Epub 2016 Nov 14.
9. Altman D, Geale K, Falconer C, Morcos E. A generic health-related quality of life instrument for assessing pelvic organ prolapse surgery: correlation with condition-specific outcome measures. Int Urogynecol J. 2018 Mar 6. doi: 10.1007/s00192-018-3587-5.
10. Khatri G, Carmel ME, Bailey AA, Foreman MR, Brewington CC, Zimmern PE, Pedrosa I. Postoperative Imaging after Surgical Repair for Pelvic Floor Dysfunction. Radiographics. 2016 Jul-Aug;36(4):1233-56.
11. Manonai J, Rostaminia G, Denson L, Shobeiri SA. Clinical and ultrasonographic study of patients presenting with transvaginal mesh complications. Neurourol Urodyn. 2016 Mar;35(3):407-11. doi: 10.1002/nau.22725. Epub 2015 Jan 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated by one of the procedures mentioned 1. Anterior TVM (Uphold™ Lite Vaginal mesh - Boston Scientific. 2. Posterior POP mesh (Pinnacle posterior - Boston Scientific or equal) 3. Y-shaped mesh via robotic assisted sacroclpopexy (Artisyn® Y-Shaped Mesh - Ethicon or equal). and 4. patients received anterior and/or posterior colporraphy i.e. native tissue repair i.e. no synthetic materials used (control group).
* All patients should have suffered prolapse symptoms before surgery such as pelvic heaviness and/or vaginal bulging, extra.
* Being able to make an informed consent on participation
* Physically and cognitively capable of participating in the examination
* No exclusion criteria fulfilled

Exclusion Criteria:

* Patients operated by different procedures t.ex. two different mesh types
* Advanced procedure in the pelvic floor such as current pelvic organ cancer (regardless of treatment)
* Other clinically relevant pelvic disorders for which surgery with other materials (not polypropylene mesh) was previously provided.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are only females previousely received surgery for female genital prolapse.
Study Population: Patients operated by one of the procedures:
  1. Anterior TVM (Uphold™ Lite Vaginal mesh - Boston Scientific.
  2. Posterior POP mesh (Pinnacle posterior - Boston Scientific or equal)
  3. Y-shaped mesh via robotic assisted sacroclpopexy (Artisyn® Y-Shaped Mesh - Ethicon or equal).
  4. patients received anterior and/or posterior colporraphy i.e. native tissue repair i.e. no synthetic materials used (control group).
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-10-21 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Detection of which mesh without being informed of previous surgery | Maximum of 10 minutes for all examination
  Without being informed of previous surgery, examiners are to separately diagnose which mesh vs no mesh
Precision of mesh detection | Maximum of 10 minutes for all examination
  Being informed of which surgery, examiners are to separately measure the midsagittal lengths of the mesh.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Morcos, MD, PhD, Principal Investigator — Karolinska Institutet - Danderyds Sjukhus (KIDS)
Locations (1):
- Division of Obstetrics and Gynecology, Department of Clinical Sciences, Karolinska Institutet Danderyd University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD is only available to the principal investigator.